CLINICAL TRIAL: NCT05678075
Title: An Educational Campaign to Stimulate Adoption of a Whole-Food Plant-Based Diet Amongst Stanford Physicians: The PLANT Study (Providers Learning About Nutrition Together)
Brief Title: The Stanford Plant-based Educational Study: Providers Learning About Nutrition Together (PLANT)
Acronym: PLANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tamiko Katsumoto, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 68145
Record Dates: First submitted 2023-01-01; First posted 2023-01-10 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Diet, Healthy
Keywords: plant-based diet; physician nutrition education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole food plant-based nutrition education (Active Comparator): Providers will receive an educational intervention on whole food plant based nutrition that will last 6 weeks.
  Interventions: Behavioral: Whole-food plant-based nutrition education
- Delayed intervention (No Intervention): Providers will receive a educational intervention on whole food plant based nutrition that will last 6 weeks.

INTERVENTIONS:
Behavioral: Whole-food plant-based nutrition education — Participants will receive an educational intervention regarding the benefits of a whole food plant-based diet and how to incorporate more plant-based foods into their diets. The intervention will last 6 weeks.
  Arms: Whole food plant-based nutrition education

SUMMARY:
More than 70% of chronic illnesses can be prevented or reversed with a whole-food, plant-based diet (WFPBD). This dietary pattern is also more sustainable for our planetary health. The majority of physicians receive fewer than 20 hours of nutrition education during the entire course of their medical training. Although many physicians are aware of the importance of diet on their well-being, they face significant barriers in following a healthy diet. Because physicians' own habits strongly influence patient health habits, the investigators theorize that physicians who eat a WFPBD themselves will be much more likely to successfully counsel their patients on nutrition and recommend a WFPBD.

The most effective methods that can be successfully used to encourage busy physicians to adopt a WFPBD have not yet been identified. Given the increasing rates of diet-related chronic illnesses, if proven effective, this study may offer a new scalable approach to encourage physicians, and ultimately their patients, to adopt a WFPBD.

The aims of this study are to:

1. Assess the impact of a multimodal 6-week educational program on WFPBD on a) change in physicians' diet type and quality, b) change in mindset about WFPBD, and c) stage of change based on the transtheoretical model of behavior change (Figure 1), compared to the delayed-intervention (control group) from baseline to week 6.
2. Assess the impact of the 6-week educational program on the development of skills and knowledge required to a) adopt a WFPBD and b) counsel patients on the same.

DETAILED DESCRIPTION:
Study overview:

This is a randomized, delayed intervention trial testing a flexible, multimodal WFPBD educational program for 6 weeks for providers at Stanford in any department.

Research Activities:

1. Screening: Interested participants will participate in a Qualtrics survey, which will determine eligibility.
2. Enrollment: If the provider expresses interest in participating, the research team will send an email that explains details about the study. A waiver of consent will be utilized given minimal risk.
3. Intervention: a 6-week multimodal educational intervention program. We will utilize a pre- and post-study survey which will include information on current dietary habits and use of Diet ID (assessment of diet type and quality). We will also assess their mindset for adopting a WFPBD. Finally, we will assess measures of motivation and confidence to adopt a WFPBD and to prescribe a WFPBD to patients. The educational program will include interactive didactic sessions, cooking classes, and weekly emails with suggested resources and activities including movies, recipes, and websites.

ELIGIBILITY:
Inclusion Criteria:

* Clinical personnel at Stanford who agree to participate in this nutritional intervention study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Diet ID score from baseline to Week 6 | 6 weeks
  Change in Diet ID score (measuring diet type and quality, on an ordinal scale of 1-10 with higher values representing better quality) will be assessed using the validated Diet ID tool
Change in mindset about WFPBD from baseline to week 6 | 6 weeks
  Change in mindset about WFPBD will be assessed using a validated survey
Change in state of change (motivation/confidence) from baseline to week 6 | 6 weeks
  Change in stage of change (motivation and confidence) will be assessed using the validated survey for transtheoretical model of behavior change

CONTACTS AND LOCATIONS:
Overall Officials: Tamiko Katsumoto, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No